CLINICAL TRIAL: NCT04848545
Title: Prenatal Exposure to Endocrine Disrupting Chemicals and Risk of Testicular Cancer in Offspring
Brief Title: Endocrine Disrupting Chemical Exposure and Testicular Cancer
Acronym: DISRUPT
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Juul, Head of Department of Growth and Reproduction, Rigshospitalet, Denmark
Other Study IDs: 1R01CA236816-01A1 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Amniotic fluid, blood serum and dried heel blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Live-born sons (with and without testicular cancer diagnosis) from a Danish pregnancy Cohort: Pregnancy cohort: Biological samples from 128,702 of pregnant women were stored for research purposes in the Danish National Biobank, in the period from 1976-2004.
  Present study: live-born sons (with/without testicular cancer ascertained via data linkage in the Danish Cancer Registry)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Prenatal maternal exposure to endocrine disrupting chemicals

SUMMARY:
DISRUPT is a Danish nested case-control study that is currently being conducted to explore the impact of prenatal exposure to endocrine disrupting chemicals on testicular cancer risk (including histological sub-groups) with emphasis on the analysis of exposure mixtures. Pregnant mothers provided serum and amniotic fluid at recruitment up to 50 years ago. By registry linkage within highly reliable national population and disease registries cancer cases and matched controls will be identified. Levels of EDCs including DDT, DDE and other organochlorine pesticides, PCBs, PBDEs, PFAS, phthalates and triclosan will be quantified in cases whose sons develop testicular cancer during 40 year follow up and compared to controls.

DETAILED DESCRIPTION:
Objectives and background Hypothesis: The central hypothesis is that testicular cancer has a fetal origin and that exposure to Endocrine Disrupting Chemicals (EDCs) plays a pivotal role in the programming of this disease via disruption of the natural in utero estrogen/androgen balance and dysregulation of the epigenetic control of gene expression within a critical masculinization time window of testicular differentiation in the developing male fetus from gestational weeks 8-14. There will be no (new) medical intervention, no new collection of biological material and no other strain on the mothers or sons who have already submitted the biological material.

Objectives: The overall objective of this proposal is to provide unique evidence relating pre-natal EDC exposure to the risk of testicular cancer in male offspring. The project will focus on exposures taking place in fetal life directly quantified using serum and amniotic fluid samples collected from mothers while they were pregnant with the young men now aged 21 to 40. Additionally, the investigators will use dried heel blood spots collected from the newborn sons within 5 days after birth. Only ten studies have investigated environmental risk factors and testicular cancer. These were small and addressed ongoing adult EDC exposure (often after diagnosis); not reflecting exposure levels at the critical time window in early life. This project will focus on exposures taking place in fetal life and hereby for the first time address the endocrine disruption hypothesis with respect to testicular cancer in a large epidemiological study. The specific aims are to investigate the risk of testicular cancer following in-utero exposure to EDCs including DDE (1,1-bis-(4-chlorophenyl)-2,2-dichloroethene) (major metabolite of DDT), perfluorinated alkyl substances, phthalates, triclosan and cotinine (nicotine metabolite). These compounds are selected due to ubiquitous environmental occurrence, detection in humans with evidence of transfer over placenta and their endocrine disruptive properties. Thus, the successful completion of this study will have an important impact on the epidemiological evidence in reproductive male health.

Background: Although a rare cancer in the general population, testicular cancer is the most common malignancy in men aged 20-40 years worldwide, representing around 60% of all cancers diagnosed for men in this age group. The incidence of this cancer has increased several folds in all industrialized during the 20th century. The reasons for this trend remain largely unknown and cannot be explained by established risk factors including cryptorchidism, Caucasian ethnicity or personal/family history of the cancer. Environmental exposures to chemicals disrupting natural in-utero hormone balance within a critical time of testicular differentiation in the developing male fetus may play a role and this is supported by the evolution of the incident rates between first and second-generation migrant populations. In addition, the large geographical variations in incidence in different European countries and the possible increase of environmental exposure to endocrine active xenobiotics within the same period in industrialized countries also support this. Given the peak incidence of this cancer in young men and the fact that testicular cancer (both seminomas and non-seminomas) is shown to develop through a common precursor -the carcinoma-in situ cells of fetal origin; the role of early exposures, during critical time windows of testicular differentiation has also been hypothesized. This is part of a hypothesis called the testicular dysgenesis syndrome, proposing a common origin of male reproductive disorders within fetal life resulting from disturbed programming of the development of male reproductive organs as a result of endocrine disruption from exogenous compounds.

Challenges and obstacles The rarity of testicular cancer in the population, the long lag time between the presumed sensitive period during fetal development and clinical appearance and the to date lack of appropriate animal models for testicular cancer have hindered the understanding of the factors involved in the development of this cancer. Therefore, there is a need for research with reliable data based on exposure assessment quantified in biological pre-natal samples, which are considered the golden standard for exposure assessment. There is an evident gap in knowledge regarding evidence to support or refute the role of EDCs in the fetal origin of testicular cancer. Based on quantification of EDC exposures in biological samples collected during pregnancy and ascertainment of outcomes in high quality, complete nationwide Danish registries, this study will provide unprecedented data on risk of testicular cancer following pre-natal exposure to EDCs.

Unique biobank (already established). All Danish women are offered a free screen for congenital diseases and chromosomal defects in offspring in the first trimester of their pregnancy, consisting of an ultrasound scan and amniotic fluid/blood sample. Samples from 128,702 of the screened pregnant women were stored for research purposes in the Danish National Biobank, in the period from 1976-2004. Within 7 days of birth all live born children born to these women had heel-blood sampled and stored as dried blood spots at the same Danish National Biobank. This heel-blood collection is part of the national Danish screening for congenital diseases.

The unique infrastructure of Danish registries. In Denmark, information on births, deaths, immigration and emigration, disease incidence, education and social conditions has been collected in nationwide registries for several decades and high-quality data with complete coverage of the whole population is available, offering great possibilities for nationwide epidemiological studies of health effects related to environmental and lifestyle exposures that are not be feasible in most other countries. In each registry persons are each identified by a unique number, called a CPR-number. This number has been given to all residents of Denmark since the establishment of the Danish Civil Registration System (CRS)in 1968 and allows accurate linkage between registries. Using this infrastructure, the investigators can identify: (i)Study participants by linking mothers that provided blood and amniotic fluid to their live-born sons that provided heel-blood at birth. Using the mother's CPR-number that is linked to her samples in the Danish National Biobank at Staten Serum Institute the investigators can trace the CPR-number of her son in the Danish Medical Birth Registry (MBR). The MBR contains information on all live-and stillbirths in Denmark since 1973, as well as information on congenital defects including cryptorchidism of the live-born sons. Further, the MBR contains information on weight, height, age and ethnicity of mother as well as the age, ethnicity and CPR-number of the father. (ii) All sons that have developed cancer in later life with accuracy and complete coverage. Using the Danish Cancer Registry (DCR), which is a population-based registry containing data on the incidence of all cancers since 1943, known for accuracy and complete coverage, the investigators will identify all cases of testicular cancer amongst the live-born sons (22 to 45 years old). (iii) Family history of testicular cancer with accuracy and complete coverage. Using the DCR and the father's CPR-number the investigators will trace family history of testicular disease, a known risk factor for testicular cancer in offspring [72]. All other cancers will be ascertained for the case-controls. Included controls are free of all cancers and cases with another cancer prior to testicular cancer onset will be excluded.

Expected scientific and public health impact of this proposal. The overall scientific contribution of the proposed project is to provide human data to scientists, enabling them to corroborate or refute whether fetal exposure to EDCs are associated with increased risk of testicular cancer in offspring. Currently there is little that pregnant women (and others) can do to avoid EDC exposures, which most often are "invisible" pollutants in food, cosmetics, indoor climate, air and water. If the study refutes associations this could ease concern and if an association is corroborated the evidence could assist governments and environmental protection agencies in introducing new policies that can protect vulnerable populations in home settings, schools and workplaces or implement education programs for pregnant women such that they can take sensible measures to reduce their exposure.

Methods The project will make use of maternal (serum, amniotic fluid) and newborn (dried heel-blood) samples stored at the Danish National Biobank (cf. biobank). Design (Nested case-control).

Three controls are matched to each case. Controls are free of any cancer and matched by maternal-and paternal-age, calendar month of blood sample, ethnicity and age and address at time of cancer diagnosis. This information along with family history of testicular cancer, history of any cancer in case-control population, and other a-priori determined potential confounding variables will be obtained from nationwide registries Exposure assessment (Fetal exposure to EDCs). Two sub-contractors will perform all chemical analyses of maternal levels of selected EDCs in bio-samples.

Metabolomics profiling. The Metabolomics Research Group at the Danish Center for Neonatal Screening at Statens Serum Institut will perform the analysis of the dried blood spot metabolome. A punch of 3.2 mm diameter of the neonatal dried blood spot of each child will be used for extraction. Using analytical and computational workflows previously introduced and applied by the group, a wide range of several thousands of endogenous as well as exogenous metabolites will be measured. Data will be preprocessed, and mass spectral features will be annotated to chemical structures using computational metabolomic workflows provided through the community-driven Global Natural Products Social Molecular networking (GNPS) platform. The resulting metabolite profiles will be used for statistical analysis to identify metabolites that are differentially expressed across cases and controls using diverse in-house algorithms in R and python. Outcome ascertainment (testicular cancer). Using the CPR-number the investigators will link the sons to the DCR to extract data on the first occurrence of testicular cancer. Controls are cancer and cryptorchidism free. Cases diagnosed with any cancer prior to testicular cancer will be excluded. The project duration is 60 months.

Statistical analysis Population. The investigators expect 175 testicular cancer cases (both seminoma and non-seminomas as these have a common fetal precursor) within this population of sons. Each case will be matched with three controls giving a total population of 700 men.

Statistical analyses. Logistic regression models will be used to estimate risk and 95% confidence intervals (CIs) relating compound concentrations with risk of testicular cancer. Analyses will be done for individual compounds, compound groups where relevant (total PFASs and total phthalates) and compound mixtures. Data will be analyzed with and without adjustment for a-priori determined potentially confounding variables including mothers BMI at time of the son's birth, history of testicular cancer and cotinine serum levels (marker of smoking) adjusted for gestational sampling week.

Metabolomicsprofiling. Overall variation in the metabolome related to testicular cancer will be assessed using multivariate statistical methods such as principal coordinates analyses and permutational multivariate analyses of variance (PERMANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Available stored maternal serum and/or maternal amniotic fluid

Exclusion Criteria:

* other cancer

Ages: 15 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In Denmark all women, in the first trimester of their pregnancy, are offered a free screen for congenital diseases and chromosomal defects in offspring. According to informed consent from 128,702 of the pregnant women screened in the period from 1976-2004, serum samples from these routine screens were stored the Danish National Biobank. In addition, all live born children (including all sons born to these women) in Denmark are sampled 7 days after birth for heel-blood. The heel blood is sampled as a nationwide screen for congenital diseases and all mothers have provided informed consent to storage. All live-born sons, born to these women will be identified using the CPR-number of each mother that provided a blood sample and extracting data from the Danish Medical Birth registry.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of testicular Cancer (ICD-10 code) | Testicular cancer is ascertained in live-born sons within the cohort, during the follow-up period (up to 50 years)
  Ascertained in adult men - Registry based on ICD-10 codes for testicular cancer (C62*)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, PhD, MD, Principal Investigator — Vækst og Reproduktion, Rigshospitalet
Locations (2):
- Denmark (2):
  - Department of Growth and Reproduction, Rigshospitalet, Copenhagen
  - EDMaRC, Rigshospitalet secton 5064, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided